CLINICAL TRIAL: NCT02451202
Title: A Comparison of Surgical Conditions Between Deep vs Moderate Neuromuscular Blockade With Rocuronium in Patients Undergoing Endolaryngeal Procedures.
Brief Title: Deep vs Moderate Neuromuscular Blockade With Rocuronium in Patients Undergoing Endolaryngeal Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Oraluxna Rodanant, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 51815
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Laryngoscopic Surgical Procedures
Keywords: "surgical conditions"; "deep neuromuscular blockade"; "deep neuromuscular paralysis"
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Neuromuscular Blockade arm (Experimental): After initial doses of 0.6 mg Rocuronium, a continuous infusion can be initiated to maintain 0 responses to train-of-four (TOF) stimulation or 1-2 responses to Post-Tetanic Count (PTC) (Deep NMB). The pump rate will vary and depends on the PTC value. The initial pump rate will be set at 0.5 mg/kg per hour. In case of a deviation from the required PTC value the pump rate can be increased or decreased. This was left to the discretion of the attending anaesthetist. Deep NMB should be maintained throughout the operation.
  The infusion of Rocuronium will be discontinued and Sugammadex will be given 4 mg/kg at the end of surgery, which is from deep NMB (PTC = 1-2).
  Interventions: Procedure: Deep Neuromuscular Blockade; Drug: Sugammadex; Drug: Rocuronium
- Moderate Neuromuscular Blockade arm (Active Comparator): After evidence of early spontaneous recovery (< 10% of control T1) from initial doses of 0.6 mg rocuronium, a continuous infusion can be initiated to maintain 1 to 2 responses to train-of-four stimulation (Moderate NMB). The initial pump rate will be set at 0.5 mg/kg per hour. In case of a deviation from the required TOF value the pump rate can be increased or decreased. This was left to the discretion of the attending anaesthesiologist. Moderate paralysis should be maintained throughout an operation.
  At the end of surgery, the infusion of Rocuronium will be discontinued and Sugammadex 2 mg/kg via bolus injections]will be administered at least reappearance of T2.
  Interventions: Procedure: Moderate Neuromuscular Blockade; Drug: Sugammadex; Drug: Rocuronium

INTERVENTIONS:
Procedure: Deep Neuromuscular Blockade — * During maintenance phase, if recovery after 1 Post-Tetanic-count (PTC) responses, a continuous infusion can be initiated to maintain deep NMB (TOF =0, PTC 1-2).
  * At the end of surgery, continuous infusion Rocuronium and Propofol are discontinued and paralysis will be simultaneously reversed by Sugammadex 4mg/kg from PTC 1-2.
  Arms: Deep Neuromuscular Blockade arm
Procedure: Moderate Neuromuscular Blockade — - During maintenance phase, if recovery at the presence of <10% of control T1 of TOF from initial doses of 0.6 mg rocuronium, a continuous infusion can be initiated to maintain TOF = 1 - 2. The initial pump rate will be set at 0.5 mg/kg per hour.
  Arms: Moderate Neuromuscular Blockade arm
Drug: Sugammadex
Drug: Rocuronium

SUMMARY:
It is unknown the impact of deep neuromuscular paralysis and using a novel agent, sugammadex as an reversal in endolaryngeal surgery.

We will conduct a clinical study aiming to compare two treatment strategies; Deep neuromuscular Blockade and moderate Neuromuscular Blockade. We hypothesize that deep NMB will offer better stillness. We will also descriptively examine if patients would be safely discharged from a recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 60 years; ASA I-III.
* Subjects have been planned for elective endolaryngeal. Procedures (Direct Laryngoscopy with laser (micro-)surgery in patients with Tis, T1, T2, supraglottis and glottis carcinoma)

Exclusion Criteria:

* Any renal impairment (CrCL < 80 ml/ min)
* Any hepatic impairment; Child Pugh A, B or C
* BMI > 30 kg m2
* Known or suspected generalized neuromuscular disorders
* Allergies to Rocuronium, Sugammadex, Sevoflurane, Propofol, fentanyl used during general anesthesia
* Hypersensitivity to the active substance or to any of the excipients
* Female patient who are pregnant and breastfeeding.
* Patient with poor Glasgow Coma Score and mental derangement who is unable to give informed consent.
* Patient with Tracheostomy tube.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oraluxna Rodanant, MD, Principal Investigator — Anesthesiology Department, Faculty of Medicine, Culalongkorn University.

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Neuromuscular Blockade Arm: After initial doses of 0.6 mg Rocuronium, a continuous infusion can be initiated to maintain 0 responses to train-of-four (TOF) stimulation or 1-2 responses to Post-Tetanic Count (PTC) (Deep NMB). The pump rate will vary and depends on the PTC value. The initial pump rate will be set at 0.5 mg/kg per hour. In case of a deviation from the required PTC value the pump rate can be increased or decreased. This was left to the discretion of the attending anaesthetist. Deep NMB should be maintained throughout the operation.
  The infusion of Rocuronium will be discontinued and Sugammadex will be given 4 mg/kg at the end of surgery, which is from deep NMB (PTC = 1-2).
  Deep Neuromuscular Blockade: - During maintenance phase, if recovery after 1 Post-Tetanic-count (PTC) responses, a continuous infusion can be initiated to maintain deep NMB (TOF =0, PTC 1-2).
  - At the end of surgery, continuous infusion Rocuronium and Propofol are discontinued and paralysis will be simultaneously reversed by
- Moderate Neuromuscular Blockade Arm: After evidence of early spontaneous recovery (< 10% of control T1) from initial doses of 0.6 mg rocuronium, a continuous infusion can be initiated to maintain 1 to 2 responses to train-of-four stimulation (Moderate NMB). The initial pump rate will be set at 0.5 mg/kg per hour. In case of a deviation from the required TOF value the pump rate can be increased or decreased. This was left to the discretion of the attending anaesthesiologist. Moderate paralysis should be maintained throughout an operation.
  At the end of surgery, the infusion of Rocuronium will be discontinued and Sugammadex 2 mg/kg via bolus injections]will be administered at least reappearance of T2.
  Moderate Neuromuscular Blockade: - During maintenance phase, if recovery at the presence of <10% of control T1 of TOF from initial doses of 0.6 mg rocuronium, a continuous infusion can be initiated to maintain TOF = 1 - 2. The initial pump rate will be set at 0.5 mg/kg per hour.
  Sugammadex
  Rocuronium
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade Arm | Moderate Neuromuscular Blockade Arm
Started | 51 | 51
Completed | 49 | 48
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade Arm | Moderate Neuromuscular Blockade Arm | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 97
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Year] | 42.31 (13.28) | 43.5 (11.78) | 43.03 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 26 | 28 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 48 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: "kg/m^2"] | 22.07 (5.15) | 23.75 (3.66) | 23.03 (4.35)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Have a Clinically Acceptable Surgical Conditions
Description: Proportion of patients who have a excellent and good surgical condition score
Time Frame: intraoperative
Measure: Number; unit: Proportion of patients
Groups:
- Deep Neuromuscular Blockade Arm: Deep Neuromuscular Blockade: - During maintenance phase, if recovery after 1 Post-Tetanic-count (PTC) responses, a continuous infusion can be initiated to maintain deep NMB (TOF =0, PTC 1-2).
  - At the end of surgery, continuous infusion Rocuronium and Propofol are discontinued and paralysis will be simultaneously reversed by Sugammadex 4mg/kg from PTC 1-2.
Arm/Group | Moderate Neuromuscular Blockade Arm | Deep Neuromuscular Blockade Arm
Number analyzed (Participants) | 48 | 49
Proportion of patients | 0.89 | 1

2. Secondary Outcome: Time to Modified Aldrete's Score ≥ 9
Description: Time from Post Anesthesia Care Unit (PACU) arrival to patients were considered fit for discharge from the PACU by Modified Aldrete's score assessment which scale range is from 0-10. Higher value represents a better outcome.
Time Frame: Minutes from Post Anesthesia Care Unit (PACU) arrival to patients were considered fit for discharge from the PACU.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Deep Neuromuscular Blockade Arm | Moderate Neuromuscular Blockade Arm
Number analyzed (Participants) | 49 | 48
Minutes | 27 [14 to 42] | 33 [18 to 48]

ADVERSE EVENTS:
Time Frame: 1 year and 9 months
Description: Adverse Event reporting description based on Clinicaltrials.gov definition.
Arm/Group | Deep Neuromuscular Blockade Arm | Moderate Neuromuscular Blockade Arm
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02451202/Prot_SAP_000.pdf